CLINICAL TRIAL: NCT00590369
Title: Negative Pressure Wound Therapy: Are All Systems Alike?
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: The Cleveland Clinic (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Nancy M. Albert PhD, RN, Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8309-c; OSR 20050803; NCT00583141 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): KCI VAC type negative pressure wound therapy device
  Interventions: Device: KCI -VAC
- 2 (Experimental): Versatile One (EZCare) negative wound therapy device
  Interventions: Device: Versatile One (EZCare)

INTERVENTIONS:
Device: KCI -VAC — Negative pressure wound therapy device
  Arms: 1
Device: Versatile One (EZCare) — Negative pressure wound therapy device
  Arms: 2

SUMMARY:
Hypotheses: (1)Wound healing during hospital stay will be equal between systems, (2)RNs will perceive the Versatile One (EZCare) system as easier to use, (3)Costs related to dressing changes will be less with Versatile one (EZCare), (4)Hospital length of stay will be equal or shorter with the Versatile One (EzCare) system, (5) Nursing time using Versatile One (EZCare) will be less than or equal to VAC system, (6) Patients will report less pain during dressing changes with Versatile One (EZCare).

DETAILED DESCRIPTION:
This is a prospective, 2 group, randomized, comparative study (sample:50; 25 in each group) that will investigate whether differences can be found in selected outcomes related to wound care, using Versatile One (EZCare)versus KCI VAC negative pressure/vacuum systems. Only wounds which currently meet criteria for such device use,and for which a physician's order has been written for the device, will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adults requiring negative pressure dressings.

Exclusion Criteria:

* Comatose
* Mentally obtunded
* Documented chronic psychiatric illness or any documented dementia significant enough to notably impair cognitive function
* Presence of Manufacturer's contraindications
* Malignancy in wound
* Untreated osteomyelitis
* Unexplored fistula
* Necrotic tissue
* Exposed blood vessels or organs
* Untreated malnutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Albert, PhD, RN, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Jan 2006-March 2008; study recruitment; study stopped due to slow enrollment rate
Groups:
- KCI VAC: KCI VAC type negative pressure wound therapy device
- Versatile One: Versatile One (EZCare)negative wound therapy device
Period: Overall Study
Arm/Group | KCI VAC | Versatile One
Started | 6 | 5
Completed | 6 (Study stopped early due to difficulty recruiting subjects) | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KCI VAC | Versatile One | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 1 | 1
Age Continuous [Median (Inter-Quartile Range); unit: years]
  median | 57 (42, 58) [35 to 58] | 49 (47, 50) [47 to 50] | 50 (42, 58) [42 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: 5 Measures of Wound Healing: Length, Width, Depth, Undermining, Tunneling
Description: differences in wound healing rate at first dressing between devices; since 5 variables were assessed via a centimeter ruler
Time Frame: first dressing change; typically within 48 hours
Measure: Median (Inter-Quartile Range); unit: centimeters
Arm/Group | KCI VAC | Versatile One
Number analyzed (Participants) | 6 | 5
centimeters
  Depth of wound | 2.5 [1.6 to 3.7] | 2.2 [2.0 to 3.0]
  Length of wound | 10.6 [6.5 to 13.8] | 16.5 [4.8 to 21]
  Width of wound | 2.75 [1.5 to 5] | 4.2 [3.5 to 5.5]
  Undermining of wound | 0 [0 to 0.5] | 0 [0 to 0]
  Tunneling of wound | 0 [0 to 0] | 0 [0 to 0]

2. Secondary Outcome: Ease of Performing Dressing Change
Description: responses to questions using a Likert scale regarding ease of dressing change; 8 characteristics; only reported is: Apply/fasten occlusive drape to secure drainage tube; scale range is 0, very difficult to do, takes a lot of time or effort or not possible to 10, simple or very easy to do
Time Frame: during hospital stay; generally 6 days
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | KCI VAC | Versatile One
Number analyzed (Participants) | 6 | 5
scores on a scale | 8.5 [7.0 to 10.0] | 6.0 [5.0 to 8.0]

3. Secondary Outcome: Ease of Providing Nursing Care
Description: nurse perception of ease of providing nursing care using a Likert-type scale; 5 items assessed. Responses to 1 item provided: Overall experience with nursing care issues related to the wound device. score range is 0, always very difficult, always a problem or not possible to 10, always easy, never or rarely a problem
Time Frame: during hospital stay; generally 6 days
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | KCI VAC | Versatile One
Number analyzed (Participants) | 6 | 5
scores on a scale | 10 [9.0 to 10.0] | 8.0 [6.0 to 10.0]

4. Secondary Outcome: Cost of Wound Care
Description: cost of device/supplies used in application and dressing changes
Time Frame: during hospital stay; generally 6 days
Measure: Mean (Standard Deviation); unit: dollars (USD)
Arm/Group | KCI VAC | Versatile One
Number analyzed (Participants) | 6 | 5
dollars (USD) | 510.18 (419.77) | 333.54 (71.69)

5. Secondary Outcome: Nursing Time
Time Frame: hospital stay; generally 6 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | KCI VAC | Versatile One
Number analyzed (Participants) | 6 | 5
minutes | 33.2 (23.8) | 38.8 (19.9)

6. Secondary Outcome: Patient Reported Pain
Description: scale of 0= no pain to 10= worst pain possible
Time Frame: at first dressing change; generally 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | KCI VAC | Versatile One
Number analyzed (Participants) | 6 | 5
units on a scale | 3.2 (3.7) | 2.4 (2.3)

ADVERSE EVENTS:
Time Frame: duration of patient enrollment- generally 6 days; serious and/or other [non-serious] adverse events were collected/assessed
Arm/Group | KCI VAC | Versatile One
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

LIMITATIONS AND CAVEATS:
small sample size; early termination; did not reach expected sample size. Single center

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No